CLINICAL TRIAL: NCT07099898
Title: Phase 3, Multicenter, Randomized, Open-label Clinical Study of GSK5764227, a B7-H3 Antibody Drug Conjugate (ADC), Compared With Topotecan in Participants With Relapsed Small Cell Lung Cancer (SCLC)
Brief Title: A Study of GSK5764227 in Participants With Relapsed Small Cell Lung Cancer (SCLC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 223674; 2025-521627-78 (EudraCT Number)
Record Dates: First submitted 2025-07-30; First posted 2025-08-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms, Lung
Keywords: Small Cell Lung Cancer (SCLC); GSK5764227; Topotecan
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK5764227 (Experimental)
  Interventions: Biological: GSK5764227
- Topotecan (Active Comparator)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Biological: GSK5764227 — GSK5764227 will be administered
  Arms: GSK5764227
Drug: Topotecan — Topotecan will be administered
  Arms: Topotecan

SUMMARY:
"In this study researchers are testing GSK5764227, a new medicine that targets specific proteins (B7-H3) on cancer cells, thereby reducing the cancers ability to grow and spread. This study specifically aims to evaluate how well GSK5764227 works in treating relapsed SCLC compared to standard treatment topotecan, by checking whether GSK5764227 makes cancers smaller or disappear completely and if it helps participants live longer. The study is also assessing whether GSK576227 is safe and tolerated well by participants compared to topotecan and provide a better understanding of the main side effects of both drugs. Participants with relapsed SCLC will be randomly divided into two groups: one group receiving GSK5764227 and the other receiving topotecan."

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Adults >18 or the minimum legal adult age at the time the informed consent form is signed
* Has histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC).
* Has received 1 prior platinum-based systemic therapy with a PD- (L)1 inhibitor with at least 2 cycles of therapy and a chemotherapy free-interval of >30 days, with documented progression
* Has at least 1 target lesion per RECIST 1.1, as determined by the investigator.
* Is capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Has an ECOG performance status of 0 or 1

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Pathological diagnosis of complex SCLC or transformed SCLC.
* Has received any prior therapy with an Antibody-drug conjugate (ADC) with a Topoisomerase-1 (TOPO1)-inhibitor payload or treatments targeting B7-H3.
* Has known sensitivity to study intervention components or excipients or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Has severe, uncontrolled or active cardiovascular disorders.
* Has clinically significant bleeding symptoms or significant bleeding tendency within 1 month prior to the first dose.
* Known active infectious diseases requiring systemic treatment or known Human immunodeficiency virus (HIV).
* Has symptomatic brain metastases or untreated progression exclusively due to brain metastasis during or after the last treatment prior to screening, evidence of leptomeningeal/meningeal/brainstem metastasis or evidence of spinal cord metastases.
* Has any evidence of current interstitial lung disease or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high dose steroids.
* Has documented Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2028-09-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 55 weeks
  ORR is defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Blinded independent central review (BICR) assessment
Overall Survival (OS) | Up to approximately 55 weeks
  OS is defined as the time from the date of randomization to the date of death by any cause

SECONDARY OUTCOMES:
ORR by investigator assessment | Up to approximately 161 weeks
  ORR is defined as the percentage of participants with a confirmed CR or confirmed PR per RECIST 1.1 by investigator assessment
Duration of Response (DoR) | Up to approximately 161 weeks
  DoR is defined as the time from the date of first documented objective response (CR or PR) per RECIST 1.1 by [investigator/BICR] assessment to the date of first documented PD per RECIST 1.1 by [investigator/BICR] assessment or death due to any cause, whichever comes first
Progression-free survival (PFS) | Up to approximately 161 weeks
  PFS is defined as the time from the date of randomization to the date of first documented Progressive disease (PD) per RECIST 1.1 by [investigator/BICR] assessment or death from any cause, whichever occurs first
Disease control rate (DCR) 12 | Up to approximately 11 weeks
  DCR12 is defined as the percentage of participants who have a Best objective response (BOR) of confirmed CR, confirmed PR, or Stable Disease (SD) after the date of randomization, per RECIST 1.1 by [investigator/BICR] assessment
Brain PFS | Up to approximately 161 weeks
  Brain PFS is defined as the time from the date of randomization to the date of first documented PD per Response assessment in neuro-oncology (RANO-BM) by Response Evaluation Criteria in Solid Tumors by blinded independent central review (RANO-BICR) assessment or death from any cause, whichever occurs first in participants with a history of brain metastasis
Brain DoR | Up to approximately 161 weeks
  Brain DoR is defined as the time from the first documented objective response (CR/PR according to RANO-BM by RANO-BICR assessment) until the time of first documentation of disease progression or death, whichever occurs first, in participants with a history of brain metastasis
Brain ORR | Up to approximately 161 weeks
  Brain ORR is defined as the percentage of participants with confirmed brain CR or confirmed brain PR per RANO-BM by RANO-BICR assessment
Brain DCR12 | Up to approximately 11 weeks
  Brain DCR12 is defined as the percentage of participants with an intracranial BOR of confirmed CR, confirmed PR or SD after the date of randomization, per RANO-BM by RANO-BICR assessment
Time to brain progression | Up to approximately 161 weeks
  Time to brain progression is defined as the time from the date of randomization to the date of first documented brain PD per RANO-BM by RANO-BICR assessment
Number of participants with Adverse events (AEs), Serious Adverse Events (SAEs) and Adverse events of special interest (AESIs) by severity | Up to approximately 161 weeks
Number of participants with AEs leading to dose modifications or study intervention discontinuation | Up to approximately 161 weeks
Number of participants with a change from baseline in vital signs | Baseline (Day -1) and up to approximately 161 weeks
  Number of participants will be assessed.
Number of participants with a change from baseline in laboratory parameters (hematology and clinical chemistry) | Baseline (Day -1) and up to approximately 161 weeks
  Number of participants will be assessed.
Number of participants with a change from baseline in cardiac function [Electrocardiogram (ECG) | Baseline (Day -1) and up to approximately 161 weeks
  Number of participants will be assessed.
Number of participants with a change from baseline in Eastern Cooperative Oncology Group (ECOG) performance status | Baseline (Day -1) and up to approximately 161 weeks
  Number of participants will be assessed.
Observed PK concentrations of GSK5764227 (conjugated antibody and small molecule payload) | Up to approximately 161 weeks
Number of participants with Antidrug antibody (ADA) or Neutralizing Antibody (NAb) | Up to approximately 161 weeks
Titers of ADA against GSK5764227 | Up to approximately 161 weeks

CONTACTS AND LOCATIONS:
Locations (51):
- Argentina (5):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Vicente López
- Australia (3):
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Nedlands, Western Australia
- Brazil (3):
  - GSK Investigational Site, CuritibaPR
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São Paulo
- Canada (3):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Vaasa, Finland
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Pylaia Thessaloniki
- GSK Investigational Site, Jerusalem, Israel
- Japan (11):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama
- Mexico (3):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
- South Korea (8):
  - GSK Investigational Site, Changwon
  - GSK Investigational Site, Cheongju Chungcheongbuk-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Gyeonggi-do
  - GSK Investigational Site, Ulsan
- GSK Investigational Site, Stockholm, Sweden
- GSK Investigational Site, Basel, Switzerland
- Turkey (Türkiye) (6):
  - GSK Investigational Site, Adana, Adana
  - GSK Investigational Site, Samsun, Atakum
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Diyarbakır
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
- United Kingdom (3):
  - GSK Investigational Site, London
  - GSK Investigational Site, Portsmouth
  - GSK Investigational Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf